CLINICAL TRIAL: NCT03547011
Title: The Efficacy of Ultrasound Guided Continuous Quadratus Lumborum Block Versus Continuous Paravertebral Block In Radical Cystectomy
Brief Title: Ultrasound Guided Continuous Quadratus Lumborum Block Versus Continuous Paravertebral Block In Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050108380 (13/6/2017)
Record Dates: First submitted 2017-12-03; First posted 2018-06-06 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Double blinded randomized study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, outcome assessors and care providers are not informed with the block type done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US guided Quadratus Lumborum block (Active Comparator): Patients will receive ultrasound guided quadratus lumborum block with 0.3 ml /kg bupivacaine 0.25% on each side with catheter insertion for maintenance doses 0.1ml/kg/hr on each side.
  Interventions: Procedure: US guided Quadratus Lumborum block
- US guided Paravertebral block. (Active Comparator): Patients will receive ultrasound guided thoracic paravertebral block with 0.3 ml/kg bupivacaine 0.25 % on each side with catheter insertion for maintenance doses 0.1 ml/kg/hr on each side.
  Interventions: Procedure: US guided Paravertebral block.

INTERVENTIONS:
Procedure: US guided Quadratus Lumborum block — Patients will receive ultrasound guided quadratus lumborum block with 0.3 ml /kg bupivacaine 0.25% on each side with catheter insertion for maintenance doses 0.1ml/kg/hr on each side.
  Arms: US guided Quadratus Lumborum block
Procedure: US guided Paravertebral block. — Patients will receive ultrasound guided thoracic paravertebral block with 0.3 ml/kg bupivacaine 0.25 % on each side with catheter insertion for maintenance doses 0.1 ml/kg/hr on each side.
  Arms: US guided Paravertebral block.

SUMMARY:
The aim of the study to compare between intraoperative and postoperative analgesic effect of ultrasound guided continuous quadratus lumborum block and continuous thoracic paravertebral block in patients operated for radical cystectomy (primary outcome). Side effects, length of hospital stay and patient satisfaction(secondary outcome).

DETAILED DESCRIPTION:
The analgesic efficacy of ultrasound guided continuous quadratus lumborum block versus continuous paravertebral block in radical cystectomy

Protocol of a thesis submitted to the Faculty of Medicine University of Alexandria In partial fulfillment of the requirements of the degree of Master of Anaesthesia And Surgical Intensive Care

By

Amr Ragheb Hieba MBBCh, Alex. Resident Alexandria University Hospitals Department of Anaesthesia and Surgical Intensive Care Faculty of Medicine University of Alexandria 2017

SUPERVISORS

Prof. Dr. Ramadan Abdelazeem Ammar Professor of Anaesthesia and Surgical Intensive care, Faculty of Medicine University of Alexandria

CO-SUPERVISOR

Dr.Mohamad Hazem Ibrahim Ahmed Sabry

Lecturer in Anaesthesia and Surgical Intensive Care, Faculty of Medicine, University of Alexandria. For his experience in regional anaesthesia.

INTRODUCTION Bladder cancer is the most common malignancy of the urinary tract and radical cystectomy remains the gold standard for management of muscle invasive disease.(1) Despite improvement in perioperative period it remains associated with a greater morbidity and more prolonged inpatient stay than other urological studies. Bowel complications particularly ileus are amongst the commonest problems that patients experience.)2,3) Pain is common after major abdominal surgeries.Uncontrolled postoperative pain increases the incidence of postoperative complications.Multimodal analgesia can improve pain control in postoperative period and reduces complications that may arise from using a single mode of analgesia.(4) Effective regional anesthesia techniques for abdominal surgery include epidural,paravertebral , transverses abdominis plane (TAP) block .multiple approaches have been used for TAP block with ultrasound guided midaxillary approach but are sometimes patchy with variable wound coverage . the use of ultrasound approach at the level of quadratus lumborum muscle is new and may provide wider spread of the local anesthetic ( T5-L1) than TAP and paravertebral blocks.(5) Studies of quadratus lumborum block show its use in postoperative analgesia in major abdominal surgery. Results have shown widespread and long-lasting analgesic effect after ovarian surgery and resulted in lower peak arterial concentrations of injected bupivacaine as compared to lateral TAPB.(6)

Similarly, thoracic paravertebral block (PVB) has been demonstrated to provide effective postoperative analgesia in patients undergoing minor and major abdominal surgery by blocking sensory innervations of the abdominal wall. PVB significantly reduces the need for supplemental opioid administration, reduces postoperative nausea and vomiting (PONV), and in some patient groups shortens length of hospital stay. Although PVB has been demonstrated to be effective in patients undergoing abdominal and thoracic surgery, its analgesic efficacy after major gynecological surgery has not, as yet, been reported .(7,8) Studies have shown that regional anesthetic technique for cancer surgery could affect recurrence or metastasis. This retrospective study suggests that paravertebral anaesthesia and analgesia for breast cancer surgery reduces the risk of recurrence or metastasis during the initial years of follow up. (9)

AIM OF THE WORK The aim of the study to compare between intraoperative and postoperative analgesic effect of ultrasound guided continuous quadratus lumborum block and continuous thoracic paravertebral block in patients operated for radical cystectomy (primary outcome). Side effects, length of hospital stay and patient satisfaction(secondary outcome).

PATIENTS

* After approval of Local Ethics Committee, and written informed consent from each patient or oral consent if illiteracy prevent a written consent, The present study will be carried out in the Urosurgery department at Alexandria Main University hospital on 60 adult patients scheduled for radical cystectomy, males and females.
* Patients will be randomly assigned into two equal groups (30 patients each) according to type of the block:

  1. Group I:

     Patients will receive ultrasound guided quadratus lumborum block with 0.3 ml /kg bupivacaine 0.25% on each side with catheter insertion for maintenance doses 0.1ml/kg/hr on each side.
  2. Group II:

Patients will receive ultrasound guided thoracic paravertebral block with 0.3 ml/kg bupivacaine 0.25 % on each side with catheter insertion for maintenance doses 0.1 ml/kg/hr on each side.

Exclusion Criteria:

* Patient refusal.
* Coagulopathy/ thrombocytopenia.
* Localized infection at the proposed site of injection.
* Inability to comprehend the scoring systems to be employed due to mental problems.
* known allergy to the drugs to be used (local anesthetics, opioids)
* Opioid tolerance/ dependence
* Back abnormalities.
* Neurological deficits

METHODS

Pre-operative assessment and preparation:

1. History taking ,
2. Clinical examination ,
3. All needed laboratory investigations. The technique ofanaesthesiawill be explained to patients.

Premedication:

All patients will be premedicated with midazolam 0.05 mg/kg IV 30 min before surgery.

Anaesthetic technique:

A multichannel monitor will be connected to the patient to display continuous electrocardiography monitoring for heart rate (beat/min) and detection of dysrhythmias, noninvasive arterial blood pressure (mmHg), respiratory rate and arterial oxygen saturation (SpO2) .

Baseline monitoring data (blood pressure, heart rate, respiratory rate and oxygen saturation) will be recorded.

Induction of anaesthesia will be carried out with fentanyl citrate (1µ/kg)i.v, propofol 2mg/kg i.v will be injected till loss of verbal communication and endotracheal intubation will be facilitated by rocuronium bromide 0.6mg/kg.

Ventilation will be maintained with Drager fabius plus ventilator as IPPV volume control.

Anaesthesia will be maintained with Isoflurane in 100% oxygen, intermittent boluses of Rocuroniun (0.1mg/kg).

Technique of QL block group After induction of general anesthesia,the patient will be positioned for lateral position to obtain appropriate view of QL and thoracic PV block.Aseptic measures will be taken by wearing sterile gown and sterile drapes .Ultrasound will be used with linear probe covered with sterile elastic sheath. Probe will be placed horizontally between the costal margin and iliac crest. The 3 muscle layer of the abdominal wall will be identified as external oblique, internal oblique , transverses abdominis muscles .The fascia surrounding transverses abdominis will be tracked until its origin, where transverses abdominis muscle merge with thoracolumbar fascia surrounding quadratus lumborum muscle .

18 G 3 inch long non stimulating echoic needle will be inserted in plane with the ultrasound probe and targeted toward fascia transversalis . Normal saline 3 ml will be used to identify the splitting of the fascia .Then injection of 0.3 ml/kg bupivacaine 0.25% in the same plane after negative aspiration.

This will be seen spreading around quadratus lumborum muscle. Echogenic catheter will be advanced 7 cm beyond the tip of the needle with minimal resistance.(10) Maintenance will be 0.1 ml\kg\hr. The procedure will be repeated on the other side after placing the patient in the opposite position.

Technique for thoracic paravertebral block After general anesthesia, the patient will be positioned to lateral position. Under strict aseptic technique, Ultrasound will be used with linear probe covered with sterile elastic sheath .Probe is applied longitudinal at level of T10.

For most of patients, the depth of field is set to 3 cm to start scanning. The transverse processes and ribs are shown as hyperechoic structures with acoustic shadowing between them.

Once the transverse processes and ribs are identified, the transducer is moved slightly cauded into the intercostals space between adjacent ribs to identify the thoracic PVS and adjoining intercostal space.

The PVS appears as a wedge shaped hypoechoic layer demarcated by the hyperechoic reflections of the pleura below and internal intercostal membrane above.

The hyperechoic line of the pleura and underlying hyperechoic air artifacts move with respiration .the goal of the technique is to insert the needle into PVS to inject 0.3ml∕kg bupivacaine 0.25% .(11) Echogenic catheter is advanced 7 cm beyond the tip of the needle with minimal resistance.

Maintenance will be 0.1ml\kg\hr. The same procedure will be repeated on the other side after placing the patient in the opposite position .

Measurements

The following parameters will be measured :

A- Hemodynamic parameters :

* Heart rate (beat per minute )
* Mean arterial blood pressure (mmHg)
* Oxygen saturation using pulse oximetry . All previous parameters will be continuously monitored and recorded at the following periods : preoperative , every 30 minutes intraoperative till the end of surgery and every 12 hrs postoperative for 3 days .

B - Intensity of postoperative pain :

Patients will be asked to quantify their pain on a visual analogue scale between 0 - 10 with (0) representing no pain and ( 10 ) representing the worst imaginable pain .(12)

It will be measured postoperative every 12hrs for 3 days .

C - Analgesic requirements :

* First request of analgesia .
* Rescue analgesia in the form of nalbuphine 0.1 mg / kg will be given when VAS score ≥4 . VAS to be assessed every 12 hrs and give rescue analgesia accordingly .
* Total dose of analgesia given .

ETHICS OF RESEARCH

Research on human or human products:

Prospective study: Informed consent will be taken from patients. In case of incompetent patients the informed consent will be taken from the guardians.

All drugs used in the research are approved by the Egyptian Ministry of Health

RESULTS Results will be put in tables. Appropriate statistical analysis test will be done.

DISCUSSION The results of the study will be discussed in view of achievement of the aim and will be compared to the other studies.

ELIGIBILITY:
Inclusion Criteria:

* • After written informed consent from each patient or oral consent if illiteracy prevent a written consent, The present study will be carried out in the Urosurgery department at Alexandria Main University hospital on 60 adult patients scheduled for radical cystectomy, males and females.

  * Patients will be randomly assigned into two equal groups (30 patients each) according to type of the block:

    1. Group I:

       Patients will receive ultrasound guided quadratus lumborum block with 0.3 ml /kg bupivacaine 0.25% on each side with catheter insertion for maintenance doses 0.1ml/kg/hr on each side.
    2. Group II:

       Patients will receive ultrasound guided thoracic paravertebral block with 0.3 ml/kg bupivacaine 0.25 % on each side with catheter insertion for maintenance doses 0.1 ml/kg/hr on each side.

       Exclusion Criteria:
  * Patient refusal.
  * Coagulopathy/ thrombocytopenia.
  * Localized infection at the proposed site of injection.
  * Inability to comprehend the scoring systems to be employed due to mental problems.
  * known allergy to the drugs to be used (local anesthetics, opioids)
  * Opioid tolerance/ dependence
  * Back abnormalities.
  * Neurological deficits.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
analgesic effect | 72 hours
  Visual Analogue Scale measure and needed postoperative analgesics.0 to 10, as 0 no pain 10 the worst pain.

SECONDARY OUTCOMES:
Side effects | 30 days
  numbers of side effects
length of hospital stay | 30 days
  Number of days in hospitals
Patient satisfaction. | 30 days
  Numbers from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria Univeristy
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data results and statistical analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Before the start till publishing the study.
Access Criteria: not public only the researchers who can access the study information.

REFERENCES:
- [Background] Arumainayagam N, McGrath J, Jefferson KP, Gillatt DA. Introduction of an enhanced recovery protocol for radical cystectomy. BJU Int. 2008 Mar;101(6):698-701. doi: 10.1111/j.1464-410X.2007.07319.x. Epub 2008 Jan 8. PMID 18190646
- [Background] Novotny V, Hakenberg OW, Wiessner D, Heberling U, Litz RJ, Oehlschlaeger S, Wirth MP. Perioperative complications of radical cystectomy in a contemporary series. Eur Urol. 2007 Feb;51(2):397-401; discussion 401-2. doi: 10.1016/j.eururo.2006.06.014. Epub 2006 Jun 27. PMID 16905242
- [Background] Bulka CM, Shotwell MS, Gupta RK, Sandberg WS, Ehrenfeld JM. Regional anesthesia, time to hospital discharge, and in-hospital mortality: a propensity score matched analysis. Reg Anesth Pain Med. 2014 Sep-Oct;39(5):381-6. doi: 10.1097/AAP.0000000000000121. PMID 25025697
- [Background] Liu SS, Wu CL. Effect of postoperative analgesia on major postoperative complications: a systematic update of the evidence. Anesth Analg. 2007 Mar;104(3):689-702. doi: 10.1213/01.ane.0000255040.71600.41. PMID 17312231
- [Background] Niraj G, Kelkar A, Jeyapalan I, Graff-Baker P, Williams O, Darbar A, Maheshwaran A, Powell R. Comparison of analgesic efficacy of subcostal transversus abdominis plane blocks with epidural analgesia following upper abdominal surgery. Anaesthesia. 2011 Jun;66(6):465-71. doi: 10.1111/j.1365-2044.2011.06700.x. Epub 2011 Apr 4. PMID 21457153
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Background] Naja Z, Ziade MF, Lonnqvist PA. Bilateral paravertebral somatic nerve block for ventral hernia repair. Eur J Anaesthesiol. 2002 Mar;19(3):197-202. doi: 10.1017/s0265021502000352. PMID 12071240
- [Background] Richardson J, Vowden P, Sabanathan S. Bilateral paravertebral analgesia for major abdominal vascular surgery: a preliminary report. Anaesthesia. 1995 Nov;50(11):995-8. doi: 10.1111/j.1365-2044.1995.tb05939.x. PMID 8678263
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- [Background] Bouzinac A, Delbos A, Mazieres M, Rontes O. [Ultrasound-guided bilateral paravertebral thoracic block in an obese patient]. Ann Fr Anesth Reanim. 2011 Feb;30(2):162-3. doi: 10.1016/j.annfar.2010.11.021. Epub 2011 Feb 1. No abstract available. French. PMID 21282032
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510